CLINICAL TRIAL: NCT01329848
Title: Using Accommodative Lag to Diagnose Accommodation Disorders
Brief Title: Accommodation Disorders
Acronym: AD
Status: Completed | Type: Observational
Sponsor: Western University of Health Sciences (Other)
Collaborators: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Principal Investigator, Christopher Chase, Professor of Optometry, Western University of Health Sciences
Other Study IDs: 1R15EY021021 (NIH)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Accommodative Insufficiency; Ill-sustained Accommodation
Keywords: Accommodation; Reading; Autorefraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- discomfort symptoms: level of discomfort symptoms while performing near work

SUMMARY:
This project will develop clinically useful, objective measurements of accommodative insufficiency and fatigue using continuous autorefraction recordings. The development of these procedures will help vision care professionals diagnose and treat accommodative anomalies.

DETAILED DESCRIPTION:
This project studies accommodative function, the ability to focus while doing near work. Visual discomfort symptoms, such as headaches, sore eyes, and blurred vision are commonly associated with prolonged reading or other near work. Researchers have long suspected accommodative dysfunction was involved but most clinical studies have failed to establish a relationship between weak accommodation and symptoms or reading impairments. Recent research, however, has found that clinical measure overestimate accommodative function and encourage the use of objective, autorefraction methods to measure and study accommodative weakness. This project will accomplish three goals. First, using autorefraction objective reliable procedures will be developed for measuring accommodative lag, the difference between the target location and where the eye is focused. Second, experiments will measure in real-time the impact of accommodative lag on reading fluency and visual discomfort systems. Third, studies will explore the role of the slow adaptive component in accommodative weakness. This work will lead to better methods for diagnosing and treating accommodative disorders.

ELIGIBILITY:
Inclusion Criteria:

* older adolescent and young adult
* skilled readers who attend school
* are skilled readers
* have heavy reading demands

Exclusion Criteria:

* Age > 30.
* Abnormal vergence system.
* Dry-eye.
* Uncorrected visual defects or significant ocular pathology.
* Learning disability or low IQ
* Medical conditions that might cause uncomfortable visual symptoms (e.g., migraine headaches, epilepsy, head trauma); sensory defects (e.g., deafness), or neurological conditions (e.g., stuttering) that could impair reading development or oral reading fluency.
* Somatosensory amplification.
* Systemic illness or medication associated with accommodative dysfunction.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Graduate students from Western University of Health Sciences
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Chase, PhD, Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Discomfort Symptoms: levels of discomfort while performing near work
Period: Overall Study
Arm/Group | Discomfort Symptoms
Started | 83
Completed | 54
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: Graduate students at WesternU
Arm/Group | Discomfort Symptoms
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 83
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 83
Conlon Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Measures visual discomfort symptoms while doing near work. 23 item survey using a 4-point rating scale (never, occasionally, often, almost always). Total raw score reported on a range from 0 to 69 with higher scores indicating more frequent symptoms.
  units on a scale | 24.4 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Accommodation Lag 5D
Description: Lag will be measured at different viewing distances and durations using autorefraction. Accommodation error refers to the difference between the distance where the target is located and where the eyes focus. Lag refers error that is under focussed; lead is error that is over focussed. This distance is measured in diopters, or 1/meter.
Time Frame: 3 week period
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Discomfort Symptoms
Number analyzed (Participants) | 54
diopters | 0.9 (0.6)

2. Secondary Outcome: Conlon Symptom Survey
Description: Measures visual discomfort symptoms while doing near work. 23 item survey using a 4-point rating scale (never, occasionally, often, almost always). Total raw score reported on a range from 0 to 69 with higher scores indicating more frequent symptoms.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Discomfort Symptoms
Number analyzed (Participants) | 54
units on a scale | 18.6 (12.7)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Changes in Visual Discomfort From Baseline: Visual discomfort while making auto-refraction recordings.
Arm/Group | Changes in Visual Discomfort From Baseline
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes